CLINICAL TRIAL: NCT05648565
Title: Effects of Radiofrequency Ablation of Posterior Nasal Nerves on Inflammatory Cytokines, Peak Nasal Inspiratory Flow, and Nasal Blood Flow in Patients With Chronic Rhinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: American Academy of Otolaryngic Allergy (Other)
Responsible Party: Principal Investigator, David Z. Allen, Resident, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-22-0899
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Results first posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Chronic Rhinitis
Keywords: radiofrequency ablation
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Radiofrequency ablation (RFA) (Experimental)
  Interventions: Device: Radiofrequency ablation (RFA)

INTERVENTIONS:
Device: Radiofrequency ablation (RFA) — The NEUROMARK device is an in-office, disposable bipolar RFA device with a treatment tip consisting of micro electrodes which delivers RF energy while monitoring appropriate tissue contact to maximize delivery to posterior nasal nerve and its variable branching. After topical anesthesia consisting of oxymetazoline and 1% lido followed by 4% lidocaine, the device will be placed in the posterior inferior turbinate under endoscopic visualization. The device will be activated per manufacturer's instructions

SUMMARY:
The purpose of this study is to assess the effectiveness of radiofrequency ablation (RFA) of the posterior nasal nerve (PNN) in chronic rhinitis (CR) patients by comparing patient reflective total nasal symptom score (rTNSS) and nasal obstruction symptom evaluation (NOSE) , peak nasal inspiratory flow (PNIF) , and levels of Type 2 cytokines pre- and post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* chronic rhinitis symptoms for at least 6 months (rhinorrhea, congestion, post-nasal drip)
* poor response to medical management that was attempted for at least 4 weeks
* a rTNSS score ≥6, as well as ≥2 for rhinorrhea, and ≥1 for congestion.

Exclusion Criteria:

* active sinusitis
* rhinitis medicamentosa
* recurrent and ongoing epistaxis
* immunodeficiency as defined by an illness or a history of sinus surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Z Allen, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiofrequency Ablation (RFA)
Started | 17
Received Intervention | 15
Completed | 13
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Radiofrequency Ablation (RFA)
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.18 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Nasal Congestion as Assessed by the Peak Nasal Inspiratory Flow (PNIF)
Description: PNIF is used to assess nasal air flow during maximal inspiration, and is reported in liters per minute.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: Liters Per Minute
Arm/Group | Radiofrequency Ablation (RFA)
Number analyzed (Participants) | 15
Liters Per Minute | 90 [66.6 to 113.4]

2. Primary Outcome: Nasal Congestion as Assessed by the Peak Nasal Inspiratory Flow (PNIF)
Description: PNIF is used to assess nasal air flow during maximal inspiration, and is reported in liters per minute
Time Frame: 4 weeks post intervention
Population: Data were not collected from 6 participants in the Radiofrequency ablation (RFA) arm.
Measure: Median (Inter-Quartile Range); unit: Liters Per Minute
Arm/Group | Radiofrequency Ablation (RFA)
Number analyzed (Participants) | 11
Liters Per Minute | 85 [46.9 to 123.1]

3. Primary Outcome: Nasal Congestion as Assessed by the Peak Nasal Inspiratory Flow (PNIF)
Description: PNIF is used to assess nasal air flow during maximal inspiration, and is reported in liters per minute
Time Frame: 12 weeks post intervention
Population: Data were not collected from 5 participants in the Radiofrequency ablation (RFA) arm.
Measure: Median (Inter-Quartile Range); unit: Liters Per Minute
Arm/Group | Radiofrequency Ablation (RFA)
Number analyzed (Participants) | 12
Liters Per Minute | 85 [58.1 to 111.9]

4. Primary Outcome: Interleukin-10 (IL-10)
Description: cytokine
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | Radiofrequency Ablation (RFA)
Number analyzed (Participants) | 15
picogram per milliliter (pg/mL) | 1.63 (4.28)

5. Secondary Outcome: Nasal Congestion as Assessed by the Reflective Total Nasal Symptom Score (rTNSS)
Description: This is a 4 item questionnaire and each is scored from 0(none) to 3(severe). The sum of the 4 times were added to generate a scale from 0 to 12, a higher number indicating more congestion
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Radiofrequency Ablation (RFA)
Number analyzed (Participants) | 15
score on a scale | 7 [2.9 to 5.1]

6. Secondary Outcome: Nasal Congestion as Assessed by the Reflective Total Nasal Symptom Score (rTNSS)
Description: as for outcome 5
Time Frame: 4 weeks post intervention
Population: Data were not collected from 6 participants in the Radiofrequency ablation (RFA) arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Radiofrequency Ablation (RFA)
Number analyzed (Participants) | 11
score on a scale | 4 [2.8 to 5.3]

7. Secondary Outcome: Nasal Congestion as Assessed by the Reflective Total Nasal Symptom Score (rTNSS)
Description: as for outcome 5
Time Frame: 12 weeks post intervention
Population: Data were not collected from 5 participants in the Radiofrequency ablation (RFA) arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Radiofrequency Ablation (RFA)
Number analyzed (Participants) | 12
score on a scale | 4 [2 to 6]

8. Secondary Outcome: Nasal Obstruction as Assessed by the Nasal Obstruction Symptom Evaluation Survey (NOSE)
Description: This is a 5 item self reported questionnaire and each is scored from 0(not a problem) - 4(severe problem). The sum of the 5 items were multiplied by 5, to generate a scale from 0 to 100, a higher score indicated more obstruction.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Radiofrequency Ablation (RFA)
Number analyzed (Participants) | 15
score on a scale | 50 [30 to 70]

9. Secondary Outcome: Nasal Obstruction as Assessed by the Nasal Obstruction Symptom Evaluation Survey (NOSE)
Description: as for outcome 8
Time Frame: 4 weeks post intervention
Population: Data were not collected from 6 participants in the Radiofrequency ablation (RFA) arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Radiofrequency Ablation (RFA)
Number analyzed (Participants) | 11
score on a scale | 10 [0 to 22.5]

10. Secondary Outcome: Nasal Obstruction as Assessed by the Nasal Obstruction Symptom Evaluation Survey (NOSE)
Description: as for outcome 8
Time Frame: 12 weeks post intervention
Population: Data were not collected from 5 participants in the Radiofrequency ablation (RFA) arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Radiofrequency Ablation (RFA)
Number analyzed (Participants) | 12
score on a scale | 17.5 [0 to 28.1]

11. Primary Outcome: Interleukin-22 (IL-22)
Description: cytokine
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | Radiofrequency Ablation (RFA)
Number analyzed (Participants) | 15
picogram per milliliter (pg/mL) | 0.45 (1.22)

12. Primary Outcome: Interleukin-10 (IL-10)
Description: cytokine
Time Frame: 12 weeks post intervention
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | Radiofrequency Ablation (RFA)
Number analyzed (Participants) | 13
picogram per milliliter (pg/mL) | 9.05 (38.06)

13. Primary Outcome: Interleukin-22 (IL-22)
Description: cytokine
Time Frame: 12 weeks post intervention
Population: cytokine
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | Radiofrequency Ablation (RFA)
Number analyzed (Participants) | 13
picogram per milliliter (pg/mL) | 0.37 (3.13)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Radiofrequency Ablation (RFA)
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 3/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiofrequency Ablation (RFA) (N=17)
Headaches (General disorders) | 3
dental infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-19): https://cdn.clinicaltrials.gov/large-docs/65/NCT05648565/Prot_SAP_000.pdf